CLINICAL TRIAL: NCT00218569
Title: Combined Treatment for Cocaine-Alcohol Dependence
Brief Title: Combined Treatment for Cocaine-Alcohol Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joy Schmitz, Professor - Psy, Behavioral Science, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-15801-1; R01DA015801 (NIH); R01-15801-1
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Alcohol Dependence; Cocaine Dependence
Keywords: Alcohol Dependence; Cocaine Dependence
MeSH Terms: conditions — Alcoholism; Cocaine-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Naltrexone
  Interventions: Drug: Naltrexone
- 2 (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — Naltrexone
  Other Names: Naltrexone 100mg/day
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to examine whether Naltrexone and cognitive behavioral therapy can be helpful in patients who want to stop using cocaine and alcohol.

DETAILED DESCRIPTION:
This is a randomized, double blind placebo-controlled trial to examine the role of Relapse Prevention (RP) and Contingency Management (CMP) combined with Naltrexone (NTX) for the treatment of cocaine-alcohol dependence. Patients will be randomly assigned to NTX (100mg/d) or placebo combined with one of two psychotherapy conditions (RP or RP +CMP). Following a standardized consent and intake procedure patients will participate in a 12-week trial with thrice weekly visits. Manual-guided RP therapy will be delivered in weekly 60-minute individual sessions. CMP will be based on cocaine-negative urine screens and negative breath alcohol tests. Follow-up assessments will be conducted at 3 and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Give informed consent
* Be able to understand the nature of the study, agree to comply with study requirements, report regularly for scheduled visits, and communicate with study personnel about adverse events and concomitant medication use
* Be between 18 and 60 years old
* Meet DSM-IV criteria for both current cocaine and alcohol dependence
* Be in acceptable health based on physical exam, lab tests, and EKG
* Have a stable living situation and the availability of at least two locators
* Be able to read and write English at the 6th grade level
* Provide a least one cocaine positive urine during intake
* If female, must agree to use contraception

Exclusion Criteria:

* History of evidence of a medical condition that would expose them to an undue risk or interfere with assessments during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, or neurologic disease as determined by the clinical judgment of the research team
* Medical condition that is contraindicated with opioid antagonists or necessitates opiate medication
* Abnormal liver function test results (both ALT and AST >3x upper limit normal or either >5x upper limit normal)
* Currently in treatment or have received treatment in the past six months for substance abuse or another psychiatric condition
* Evidence of a Axis I disorder that will interfere with the course of the trial, including but not limited to current Major Depressive Disorder, Bipolar Disorder, Panic Disorder, Schizophrenia, Bulimia nervosa or Anorexia, and Post-traumatic stress disorder as determined by the clinical judgment of the research team
* Participating in 12 step meetings more than twice weekly
* Opiate abuse or dependence in the last five years or used opiates, barbiturates, benzodiazepines in the last thirty days
* Current dependence on any psychoactive disorder other than nicotine
* Impending incarceration
* Condition of probation or parole requiring reports of drug use to officers of the court
* Women of child bearing potential must not be pregnant/lactating or unwilling to use an acceptable contraceptive method
* Plans to move from the Houston area within the next three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2003-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Urine toxicology for cocaine | 12 weeks of study

CONTACTS AND LOCATIONS:
Overall Officials: Joy Schmitz, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Sci Cntr Houston, Houston, Texas, United States